CLINICAL TRIAL: NCT04311307
Title: Endogenous Glucose Production in Subjects With Glycogen Storage Disease Type Ia Estimated by a Single Oral Dose of Stable Isotopes: an Investigator-initiated Human Pilot Study
Brief Title: Endogenous Glucose Production in Patients With Glycogen Storage Disease Type Ia
Acronym: ENGLUPRO GSDIa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Principal Investigator, Terry G.J. Derks, MD, PhD, Principal Investigator, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL73191.042.20
Record Dates: First submitted 2020-02-25; First posted 2020-03-17 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Glycogen Storage Disease Type IA
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): GSDIa patients
  Interventions: Biological: [6,6-2H2]glucose
- Controls (Active Comparator): Healthy volunteers
  Interventions: Biological: [6,6-2H2]glucose

INTERVENTIONS:
Biological: [6,6-2H2]glucose — Each subject will be administered two oral [6,6-2H2]glucose loads (pre-prandial, fed) in the hospital setting and one oral [6,6-2H2]glucose load at home setting (random time). Capillary blood samples will be collected on filter paper 10 times at specific time points after each oral [6,6-2H2]glucose load.

SUMMARY:
Glycogen storage disease type Ia (GSDIa) subjects retain a limited capacity for endogenous glucose production (EGP). To date, the origin of residual EGP in GSDIa patients is unknown. Either increased glycogen debranching or lysosomal glycogen breakdown can account for residual EGP in GSDIa.

Innovative treatments for GSDIa (e.g. AAV8-mediated gene therapy and mRNA therapy) are being developed.Therefore, longitudinal minimally-invasive monitoring of outcomes after therapeutic interventions in GSD Ia subjects becomes warranted.

The primary objective is to test the feasibility of EGP quantification in adult GSDIa subjects by stable isotopes after a single oral [6,6-2H2]glucose dose. Secondary objectives are to compare EGP assessed by a single oral [6,6-2H2]glucose dose (a) in GSDIa patients versus matched healthy participants, (b) among GSDIa patients, (c) in the pre-prandial state versus the fed state, (d) in the controlled hospital setting versus the home setting. Data collected from the continuous glucose monitoring data will also be compared

DETAILED DESCRIPTION:
Study design: An investigator-initiated human pilot-study. Study population: Ten adult subjects with GSDIa and ten age and gender-matched healthy subjects.

Interventions: Three experiments will be performed for each subject. During the first in hospital experiment, two oral D-[6,6-2H2]glucose loads will be performed 2 hours before breakfast and at lunchtime, respectively. The third oral D-[6,6-2H2]glucose load will be performed at home (random time). Capillary blood samples will be collected on filter paper at specific time points after each oral D-[6,6-2H2]glucose load. During the experiments, subjects will be monitored by subcutaneous continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis should be confirmed by G6PC mutation analysis
* Age above 16 years
* Stable medical condition before the start of the test procedures

Exclusion Criteria:

* Age < 16 years
* Intercurrent illness
* Recent history of hospitalization due to hypoglycemia
* Pregnancy
* History suggestive of diabetes or fasting intolerance
* First grade family member with a confirmed diagnosis associated with fasting intolerance

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
[6,6-2H2]glucose concentration in GSDIa patients | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
  Endogenous glucose production (EGP) in GSDIa will be assessed through minimal model calculation

SECONDARY OUTCOMES:
[6,6-2H2]glucose concentration in GSDIa patients and matched healthy participants | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
[6,6-2H2]glucose concentration in severe and attenuated GSDIa patients | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
[6,6-2H2]glucose concentration in the pre-prandial state versus the fed state in GSDIa patients | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
[6,6-2H2]glucose concentration in the pre-prandial state versus the fed state in healthy participants | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
[6,6-2H2]glucose concentration in the controlled hospital setting versus the home setting in GSDIa patients | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load
[6,6-2H2]glucose concentration in the controlled hospital setting versus the home setting in healthy participants | every 10 minutes within the first hour as well as 75, 90 and 120 minutes after the oral load

CONTACTS AND LOCATIONS:
Locations (1):
- University of Groningen, UMC Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Rossi A, Venema A, Haarsma P, Feldbrugge L, Burghard R, Rodriguez-Buritica D, Parenti G, Oosterveer MH, Derks TGJ. A Prospective Study on Continuous Glucose Monitoring in Glycogen Storage Disease Type Ia: Toward Glycemic Targets. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3612-e3623. doi: 10.1210/clinem/dgac411. PMID 35786777